CLINICAL TRIAL: NCT06021275
Title: Microneedling With Regular Insulin Versus Microneedling Alone in Treatment of Atrophic Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dalia Ibrahim Halwag, Lecturer and Consultant of Dermatology, Venereology and Andrology, Faculty of Medicine, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Scar 1
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Scars; Insulin
Keywords: Insulin; scars
MeSH Terms: conditions — Cicatrix; Insulin Resistance | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedling with topical application of regular insulin (Active Comparator)
  Interventions: Other: Microneedling with topical application of regular insulin
- Microneedling only (Active Comparator)
  Interventions: Other: Microneedling with topical application of saline

INTERVENTIONS:
Other: Microneedling with topical application of regular insulin — Microneeling preformed onto the scar In one group insulin will be applied while saline will be used in the second group
  Arms: Microneedling with topical application of regular insulin
Other: Microneedling with topical application of saline — Microneeling preformed onto the scar In one group insulin will be applied while saline will be used in the second group
  Arms: Microneedling only

SUMMARY:
Recently, few studies have attempted to test the regenerative effects of human insulin application by microneedling on atrophic scars versus other topical preparations. However, the scars were limited etiologically to acne scars. In addition, a lack of inclusion of a control group instead of comparing topical preparations with insulin was also a limitation to these studies. A control group consisting of microneedling alone would have served as a better comparison in order to determine whether the effects of microneedling are augmented by topical protein-rich preparations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 12 to 60 years
2. Atrophic scars (traumatic or surgical)
3. Completely healed scars

Exclusion Criteria:

1. Patients with a tendency or history of hypertrophic or keloidal scars
2. Patients who received treatment for their scar in the past 3 months
3. Diabetic patients or those with a history of Dysglycemia
4. Pregnant, or lactating females
5. Patients with active infection at the site of scar
6. Patients currently receiving isotretinoin treatment or in the past month

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in Scar | 4 months
  According the different scar assessment scores (e.g.POSAS score - The Patient and Observer Scar Assessment Scale score, range from 6 to 60, the higher the score the worse the scar, lowering in the score denotes improvement )

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Study protocol after finishing all the research and publishing the research